CLINICAL TRIAL: NCT04054999
Title: The Efficacy of Intravenous Hydroxocobalamin Versus Methylene Blue as Treatment for Intraoperative Vasoplegic Syndrome in Liver Transplant Patients
Brief Title: Methylene Blue vs Cyanokit for Intraoperative Vasoplegic Syndrome in Liver Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sher-Lu Pai, Consultant in Anesthesia, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-006247
Record Dates: First submitted 2019-08-12; First posted 2019-08-13 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Vasoplegic Syndrome; Liver Transplant; Complications
Keywords: hydroxocobalamin; methylene blue
MeSH Terms: conditions — Vasoplegia | interventions — Hydroxocobalamin; Methylene Blue

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, pilot study to describe the efficacy of hydroxocobalamin vs methylene blue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyanokit (Experimental): Single dose intraoperatively of Hydroxocobalamin (Cyanokit): 5g IV infusion over 15 minutes
  Interventions: Drug: Hydroxocobalamin
- Methylene Blue (Active Comparator): Single dose intraoperatively of Methylene blue (PROVAYBLUETM), 2 mg/kg IV bolus administered over 15 minutes
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Hydroxocobalamin — Hydroxocobalamin (Cyanokit): 5g IV infusion over 15 minutes
  Arms: Cyanokit
Drug: Methylene Blue — Methylene blue (PROVAYBLUETM), 2 mg/kg IV bolus administered over 15 minutes
  Arms: Methylene Blue

SUMMARY:
This study will evaluate if Hydroxocobalamin may be a new and possibly superior treatment for refractory vasoplegic syndrome during liver transplant surgery.

ELIGIBILITY:
* Patients scheduled to undergo liver transplantation
* Patients able to read and understand consent document (if patient is unable to provide an informed consent, the Legally Authorized Representative will be ask to consent on behalf of the patient).
* SVR lower than 500 dynes-sec/cm-5 intraoperatively (this criterion must be met after consent intraoperatively)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sher-Lu Pai, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyanokit | Methylene Blue
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyanokit | Methylene Blue | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Median (Full Range); unit: years] | 65 [39 to 71] | 59 [44 to 69] | 65 [39 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Systemic Vascular Resistance (SVR)
Description: SVR refers to the resistance to blood flow offered by all of the systemic vasculature, excluding the pulmonary vasculature. Measured during surgery at 15, 30, 60, 90 and 120 minutes after initiation of treatment.
Time Frame: 15, 30, 60, 90 and 120 minutes after initiation of treatment
Population: Data was not collected nor analyzed at all for one participant in the Methylene Blue arm. The number of participants analyzed at each time point differs due to some participants completing their surgery earlier than others. Those participants were out of the surgical room by those time points and data was not collected nor analyzed.
Measure: Median (Full Range); unit: dyne*sec/cm^5
Arm/Group | Cyanokit | Methylene Blue
Number analyzed (Participants) | 9 | 9
dyne*sec/cm^5
  15 minutes | 480 [350 to 850] | 410 [380 to 570]
  30 minutes: number analyzed (Participants) | 8 | 9
  30 minutes | 588 [330 to 770] | 420 [310 to 760]
  60 minutes: number analyzed (Participants) | 6 | 8
  60 minutes | 650 [390 to 1170] | 480 [300 to 940]
  90 minutes: number analyzed (Participants) | 3 | 6
  90 minutes | 571 [430 to 990] | 530 [330 to 610]
  120 minutes: number analyzed (Participants) | 3 | 3
  120 minutes | 543 [440 to 1060] | 415 [340 to 670]

2. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure (top number of blood pressure reading). Measured during surgery at 15, 30, 60, 90 and 120 minutes after initiation of treatment.
Time Frame: 15, 30, 60, 90 and 120 minutes after initiation of treatment
Population: The number of participants analyzed at each time point differs due to some participants completing their surgery earlier than others. Those participants were out of the surgical room by those time points and data was not collected nor analyzed.
Measure: Median (Full Range); unit: Millimeters of Mercury
Arm/Group | Cyanokit | Methylene Blue
Number analyzed (Participants) | 9 | 10
Millimeters of Mercury
  15 minutes | 109 [96 to 130] | 110 [63 to 120]
  30 minutes | 113 [97 to 147] | 101 [87 to 130]
  60 minutes | 120 [95 to 158] | 111 [92 to 145]
  90 minutes: number analyzed (Participants) | 8 | 9
  90 minutes | 129 [104 to 152] | 111 [90 to 162]
  120 minutes: number analyzed (Participants) | 7 | 9
  120 minutes | 116 [83 to 149] | 109 [101 to 161]

3. Primary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure (bottom number of blood pressure reading). Measured during surgery at 15, 30, 60, 90 and 120 minutes after initiation of treatment.
Time Frame: 15, 30, 60, 90 and 120 minutes after initiation of treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: Millimeters of Mercury
Arm/Group | Cyanokit | Methylene Blue
Number analyzed (Participants) | 9 | 10
Millimeters of Mercury
  15 minutes | 58 [40 to 66] | 55 [39 to 62]
  30 minutes | 57 [43 to 72] | 55 [41 to 68]
  60 minutes | 61 [39 to 73] | 55 [47 to 78]
  90 minutes: number analyzed (Participants) | 8 | 9
  90 minutes | 60 [42 to 72] | 57 [50 to 70]
  120 minutes: number analyzed (Participants) | 7 | 9
  120 minutes | 59 [47 to 78] | 57 [49 to 98]

4. Primary Outcome: Vasopressin
Description: Vasopressin as measured by the total amount of vasopressors administered. Measured at 15, 30, 60, 90 and 120 minutes after initiation of treatment.
Time Frame: 15, 30, 60, 90 and 120 minutes after initiation of treatment
Measure: Median (Full Range); unit: milli-units/kg/min
Arm/Group | Cyanokit | Methylene Blue
Number analyzed (Participants) | 9 | 10
milli-units/kg/min
  15 minutes | 0.04 [0.00 to 0.17] | 0.04 [0.00 to 3.71]
  30 minutes | 0.04 [0.00 to 0.13] | 0.04 [0.00 to 3.37]
  60 minutes | 0.00 [0.00 to 0.13] | 0.02 [0.00 to 0.37]
  90 minutes | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 0.37]
  120 minutes | 0.00 [0.00 to 0.11] | 0.00 [0.00 to 0.31]

5. Secondary Outcome: Post-operative Intensive Care Unit (ICU) Length of Stay
Description: Total number of days subjects were admitted to the ICU
Time Frame: Up to 30 days after surgery
Measure: Median (Full Range); unit: days
Arm/Group | Cyanokit | Methylene Blue
Number analyzed (Participants) | 9 | 10
days | 1 [0 to 20] | 0 [0 to 4]

6. Secondary Outcome: Hospital Length of Stay
Description: Total number of days subjects were admitted to the hospital
Time Frame: Up to 30 days after surgery
Measure: Median (Full Range); unit: days
Arm/Group | Cyanokit | Methylene Blue
Number analyzed (Participants) | 9 | 10
days | 7 [5 to 56] | 7 [0 to 12]

7. Secondary Outcome: Post-operative Complications
Description: The number of subjects to experience a death, cardiopulmonary event, Acute Kidney injury (AKI), Myocardial infarctions (MI), Stroke or Surgical and medical procedures - Other.
Time Frame: Up to 30 days after surgery
Measure: Number; unit: participants
Arm/Group | Cyanokit | Methylene Blue
Number analyzed (Participants) | 9 | 10
participants
  Death | 1 | 1
  Cardiopulmonary Event | 0 | 1
  AKI | 0 | 0
  MI | 0 | 0
  Stroke | 0 | 0
  Surgical and medical procedures - Other. | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline until hospital discharge, approximately two months.
Arm/Group | Cyanokit | Methylene Blue
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 1/9 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyanokit (N=9) | Methylene Blue (N=10)
Cardiopulmonary event (Cardiac disorders) | 0 | 1
Surgical and medical procedures - Other. (Surgical and medical procedures) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT04054999/Prot_SAP_000.pdf